CLINICAL TRIAL: NCT02847650
Title: A 15-WEEK, PHASE 2, DOUBLE BLIND, RANDOMIZED, PLACEBO-CONTROLLED, FLEXIBLE DOSE STUDY TO INVESTIGATE THE EFFICACY, SAFETY AND TOLERABILITY OF PF-06649751 IN SUBJECTS WITH EARLY STAGE PARKINSON'S DISEASE
Brief Title: Efficacy, Safety and Tolerability of PF-06649751 in Parkinson's Disease Patients at Early Stage of the Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study B7601011 was terminated on 29 Jan 2018 due to lack of efficacy in moderate/advanced Parkinson's disease.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: B7601011; 2016-001575-71 (EudraCT Number)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
Keywords: Early Parkinson Disease; Phase 2
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06649751 (Experimental)
  Interventions: Drug: PF-06649751

INTERVENTIONS:
Drug: Placebo
  Other Names: oral tablet once daily
  Arms: Placebo
Drug: PF-06649751
  Other Names: flexible dose oral tablet once daily
  Arms: PF-06649751

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of PF-06649751 in Parkinson's disease patients at early stage of the disease.

DETAILED DESCRIPTION:
The B7601011 study has a randomized, double-blind, placebo-controlled parallel group design. Approximately 88 subjects will be randomized to 2 treatment groups. Each subject will participate in the study for approximately 23 weeks including a 30 day screening period, 15 week double blind treatment period, and an approximately 28 day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential and/or male subjects
* Clinical diagnosis of Parkinson's disease.
* Parkinson's Disease Hoehn & Yahr Stage I-III inclusive
* Treatment naïve or history of prior incidental treatment with dopaminergic agents for no more than 28 days
* Able to refrain from any Parkinson's disease medication not permitted by the protocol.

Exclusion Criteria:

* History or presence of atypical Parkinsonian syndrome.
* Severe acute or chronic medical or psychiatric condition or cognitive impairment or laboratory abnormality.
* Any condition possibly affecting drug absorption.
* Participation in other studies involving investigational drug(s), or treatment with any investigational drug within 30 days.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (20):
  - St Joseph's Hospital and Medical Center, Barrow Neurology Clinics, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - University of South Florida Faculty Office Building, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - University of South Florida Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Asheville Neurology Specialists PA, Asheville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Gardner-McMaster Parkinson Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - AS Clinical Research Consultants of North Texas, PLLC, Greenville, Texas
  - Baylor College of Medicine, Houston, Texas
  - Sentara Neurology Specialists, Virginia Beach, Virginia
- France (8):
  - Hopital Henri Mondor, Créteil
  - Hôpital Henri Mondor, Créteil
  - CHU de Grenoble Alpes, Grenoble
  - CHU Grenoble Alpes, La Tronche
  - Hospital de La Timone, Marseille
  - Hospital La Timone, Marseille
  - Hopital Pitie Salpetriere, Paris
  - Hopital Pitie-Salpetriere, Paris
- Germany (7):
  - St. Josef Hospital GmbH, Bochum, North Rhine-Westphalia
  - Praxis Oehlwein Outpatient clinic for PD, DBS, Movement Disorders, Gera
  - Klinik Haag i. OB, Haag I. OB
  - Paracelsus-Elena-Klinik Kassel, Kassel
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - University hospital Tuebingen, Tübingen
  - Universitaetsklinik Ulm, Ulm
- Israel (2):
  - Edith Wolfson Medical Center, Holon
  - Pharmacy, Edith Wolfson Medical Center, Holon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Riesenberg R, Werth J, Zhang Y, Duvvuri S, Gray D. PF-06649751 efficacy and safety in early Parkinson's disease: a randomized, placebo-controlled trial. Ther Adv Neurol Disord. 2020 Mar 6;13:1756286420911296. doi: 10.1177/1756286420911296. eCollection 2020. PMID 32201505
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7601011

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06649751: Eligible participants were up-titrated in a double-blind fashion to an optimal dose level of PF-06649751 according to a flexible dose titration scheme (from 0.25 mg to 15 mg once daily [QD]). The 15-week treatment period included 9 weeks of dose optimization and 6 weeks of stable dosing. Blinded PF-06649751 was provided as tablets for oral administration in the outpatient setting (each morning, daily for the duration of the treatment period). Reaching of the maximum allowed dose level (15 mg) was not mandatory; participants might achieve a satisfactory clinical response at a lower dose level. There was an additional follow-up period of 28 days following discontinuation of PF-06649751.
- Placebo: Matching placebo tablet for QD dosing in the 15-week double-blind treatment period. There was an additional follow-up period of 28 days following discontinuation of placebo.
Period: Overall Study
Arm/Group | PF-06649751 | Placebo
Started | 29 | 28
Completed | 25 | 22
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06649751 | Placebo | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.76 (8.34) | 63.36 (9.16) | 64.07 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 20 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 28 | 25 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Total Score at Week 15
Description: MDS-UPDRS Part III was used to assess the motor signs of Parkinson's disease. It was comprised of 33 sub-scores based on 18 items, several with right, left or other body distribution scores. Each question was anchored with 5 responses that were linked to commonly accepted clinical terms: 0=normal, 1=slight, 2=mild, 3=moderate, and 4=severe. The MDS-UPDRS Part III total score range is 0-132. Higher score indicates more severe motor signs of Parkinson's disease. A negative change from baseline represents an improvement in motor function.
Time Frame: Baseline (Day -1/randomization), Week 15
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo) and had a baseline and Week 15 MDS-UPDRS score Part III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 25 | 22
units on a scale | -9.0 (1.54) | -4.3 (1.65)
Statistical Analysis 1: Comparison: PF-06649751 vs Placebo; Test type: Other; p = 0.0407, Mixed Models Analysis; Least Squares Mean Difference = -4.8, 90% CI 2-sided [-8.6 to -1.0], Standard Error of Mean 2.26

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: From first dose of study treatment up to 28 days after last dose (up to Day 133)
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 29 | 28
Participants
  AEs | 25 | 18
  SAEs | 1 | 0

3. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following safety laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, absolute total neutrophils, absolute eosinophils, absolute basophils, absolute monocytes, and absolute lymphocytes); chemistry (blood urea nitrogen/urea and creatinine, glucose , calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, alkaline phosphatase, uric acid, albumin, total protein); urinalysis (pH, qualitative glucose, qualitative protein, qualitative blood, ketones, nitrites, leukocyte esterase, urine bilirubin, urobilinogen, urine creatinine, microscopy, and specific gravity).
Time Frame: Baseline (Day -1/randomization) up to Day 119 follow-up visit
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo) and had at least 1 observation of the given laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 28 | 28
Participants | 19 | 19

4. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Categorical Summarization and Orthostatic Hypotension Criteria
Description: Vital signs categorical summarization criteria: 1) supine and standing systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine and standing diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) standing pulse rate <40 or >140 bpm; 5) maximum change from baseline (increase or decrease) in supine and standing DBP greater than or equal to (>=) 20 mmHg; 6) maximum change from baseline (increase or decrease) in supine and standing SBP >=30 mmHg. Orthostatic hypotension criterion was defined as a decrease of >=20 mmHg for SBP or >=10 mmHg for DBP 2 minutes after standing from a supine position.
Time Frame: Baseline (Day -1/randomization) up to Day 119 follow-up visit
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 29 | 28
Participants
  Supine SBP <90 mmHg | 0 | 0
  Standing SBP <90 mmHg | 0 | 0
  Supine DBP <50 mmHg | 0 | 0
  Standing DBP <50 mmHg | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0
  Standing pulse rate <40 bpm | 0 | 0
  Standing pulse rate >140 bpm | 0 | 0
  Maximum increase in standing DBP >=20 mmHg | 0 | 0
  Maximum increase in standing SBP >=30 mmHg | 0 | 0
  Maximum increase in supine DBP >=20 mmHg | 0 | 1
  Maximum increase in supine SBP >=30 mmHg | 0 | 3
  Maximum decrease in standing DBP >=20 mmHg | 8 | 2
  Maximum decrease in standing SBP >=30 mmHg | 4 | 1
  Maximum decrease in supine DBP >=20 mmHg | 9 | 1
  Maximum decrease in supine SBP >=30 mmHg | 5 | 0
  SBP postural difference(supine-standing) >=20mmHg | 1 | 2
  DBP postural difference(supine-standing) >=10mmHg | 3 | 1

5. Secondary Outcome: Number of Participants Meeting the Categorical Summarization Criteria for Electrocardiogram (ECG) Parameters
Description: ECG categorical summarization criteria: 1) QRS duration (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): >=140 milliseconds (msec), >=50% increase from baseline; 2) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): >=300 msec, >=25% increase when baseline is > 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec; 3) QT interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole): absolute value of >=500 msec; 4) QTcF interval (QT corrected for heart rate using Fridericia's formula): absolute value of 450 to <480 msec, 480 to <500 msec, >=500 msec; an increase from baseline of 30 to <60 msec or >=60 msec.
Time Frame: Baseline (Day -1/randomization) up to Day 119 follow-up visit
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo). "Number Analyzed" represents the number of participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 29 | 28
Participants
  PR interval >=300 msec: number analyzed (Participants) | 28 | 28
  PR interval >=300 msec | 0 | 0
  QRS duration >=140 msec | 0 | 0
  QT interval >=500 msec | 0 | 0
  QTcF interval >=450 msec to <480 msec | 0 | 0
  QTcF interval >=480 msec to <500 msec | 0 | 0
  QTcF interval >=500 msec | 0 | 0
  Percent increase in PR interval >=25/50%: number analyzed (Participants) | 28 | 28
  Percent increase in PR interval >=25/50% | 0 | 0
  Percent increase in QRS duration >=50% | 0 | 0
  Increase in QTcF interval >=30 msec to <60 msec | 1 | 2
  Increase in QTcF interval >=60 msec | 0 | 0

6. Secondary Outcome: Number of Participants With Worsening and New Onset Suicidality as Assessed by Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS responses were mapped to the Columbia Classification Algorithm of Suicide Assessment (C-CASA). Participants with new onset suicidality were those without suicidal ideation and behavior at baseline and reported any suicidal behavior or ideation post-baseline as assessed by C-CASA code mapped from C-SSRS data. Participants with worsening suicidality were those who moved to a lower numbered C-CASA category than was reported at baseline.
Time Frame: Baseline (Day -1/randomization) up to Day 119 follow-up visit
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 29 | 28
Participants
  Worsening suicidality | 0 | 0
  New onset suicidality | 1 | 0

7. Secondary Outcome: Change From Baseline in Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease - Rating Scale (QUIP-RS) Total Score at Days 35, 63, and 105
Description: The QUIP-RS has 4 primary questions pertaining to commonly reported thoughts, urges/desires, and behaviors associated with impulsive-compulsive disorder , each applied to the 4 impulsive-compulsive disorders (compulsive gambling, buying, eating, and sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). Each question is anchored with the following 5 responses: Never (0), Rarely (1), Sometimes (2), Often (3), and Very Often (4). The scoring range for each item (ie, disorder) is 0-16. The QUIP-RS total score range is 0-64. Higher score indicates a greater level of the impulsive compulsive disorder.
Time Frame: Baseline (Day -1 or randomization); Days 35, 63, 105
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo). "Number Analyzed" = Participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 29 | 28
units on a scale
  Change from baseline at Day 35: number analyzed (Participants) | 28 | 28
  Change from baseline at Day 35 | 0.2 (5.23) | 1.9 (9.49)
  Change from baseline at Day 63: number analyzed (Participants) | 27 | 24
  Change from baseline at Day 63 | -1.1 (5.99) | 1.1 (9.02)
  Change from baseline at Day 105: number analyzed (Participants) | 26 | 22
  Change from baseline at Day 105 | -1.6 (4.54) | -0.2 (5.38)

8. Secondary Outcome: Total Physician Withdrawal Checklist (PWC-20) Score
Description: The PWC-20 is a 20-item reliable and sensitive instrument for the assessment of benzodiazepine-like discontinuation symptoms. The total PWC-20 score is the sum of 20 item scores and ranges between 0 and 60. The higher score indicates more frequent/severe symptoms.
Time Frame: Day 119
Population: All participants who received at least 1 dose of study treatment (PF-06649751 or placebo) and had PWC-20 evaluation.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PF-06649751 | Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | 1.50 [0 to 12.00] | 1.00 [0 to 11.00]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 28 days after last dose (up to Day 133)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06649751 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/28
Other Adverse Events (participants affected / at risk) | 22/29 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06649751 (N=29) | Placebo (N=28)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06649751 (N=29) | Placebo (N=28)
Dry mouth (Gastrointestinal disorders) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | 2 (2)
Fatigue (General disorders) | 3 (4) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dystonia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1)
Tremor (Nervous system disorders) | 4 (5) | 2 (5)
Abnormal dreams (Psychiatric disorders) | 2 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor due to a companion study, B7601003 (NCT02687542; a dose ranging, Phase 2b study in motor fluctuators) meeting futility criteria at Interim Analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02847650/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT02847650/SAP_001.pdf